CLINICAL TRIAL: NCT05614635
Title: Prospective, Multicenter, Observational cLinical triAl Measuring Safety and Technical Performance of plAstalgin and Plastalgin Fast in Patients Requiring a Dental Impression
Brief Title: Safety and Technical Performance of Plastalgin and Plastalgin Fast in Patients Requiring a Dental Impression
Status: Completed | Type: Observational
Sponsor: Septodont (Industry)
Responsible Party: Sponsor
Other Study IDs: PLAS 2022-02; 2022-A00882-41 (Other: BRC Identification number)
Record Dates: First submitted 2022-10-24; First posted 2022-11-14 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Dental Malocclusion; Edentulous Mouth; Dental Misalignment
Keywords: Fabrication of prosthesis; Alginate Dental Impression
MeSH Terms: conditions — Malocclusion; Mouth, Edentulous

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Plastalgin and Plastalgin Fast — Plastalgin and Plastalgin Fast are potassium alginate-based powders designed for dental impression. The powder is mixed with water to obtain an impression material paste, used to imprint the teeth and mouth of the patient. The product is available under two presentations: Plastalgin and Plastalgin Fast. Plastalgin Fast has a shorter mixing time.

SUMMARY:
The aim of this study is to gather clinical data related to the use of Plastalgin and Plastalgin Fast, in order to comply with the new medical device regulation. The target population for this study is the same as the intended population specified in the study device's instructions for use: children from 5 years old and adults.

Collection, recording, and reporting of data will be accurate and will ensure the privacy, health, and welfare of participating patients during and after the study

ELIGIBILITY:
Inclusion Criteria:

* Patient fulfilling all the following criteria is eligible for the clinical investigation:
* Male or female patient ≥ 5 years of age.
* Indication of dental impressions for the fabrication of prosthesis such as mouth guards and trays, total or partial dentures, and fixed prosthesis (crowns, bridges, dental veneers).
* Total or partially edentulous patient or patient with disocclusion or patient with misalignment.
* Patient affiliated or beneficiary of a social security system.
* Written informed consent must be obtained before any study-related assessment is performed.

Exclusion Criteria:

* The presence of any of the following exclusion criteria will lead to the exclusion of the patient:
* Inability to comply with study procedures.
* Patient opposing the processing of their data.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population for this study is the same as the intended population specified in the study device's instructions for use: children from 5 years old and adults.
  Minors are eligible to participate in the study. Other vulnerable patients can be included in the study as there is no additional risk for this population.
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Anatomical reproductibility of the dental impression with Plastalgin and Plastalgin Fast. | Immediately after the procedure.
  Dentist's opinion through a questionnaire completed by the dentist

SECONDARY OUTCOMES:
Number of impressions needed per patient | Immediately after the procedure.
  Number of impressions needed per patient to make a quality impression.
Setting time of Plastalgin and Plastalgin Fast | During the procedure.
  Measure of the setting time by the dentist at each use of Plastalgin and Plastalgin Fast
Rate of adverse events | During and immediately after the procedure.
  Cumulative number of adverse events and serious adverse events
Rate of device-related adverse event | During and immediately after the procedure.
  Cumulative number of adverse events and serious adverse events related to Plastalgin or Plastalgin Fast

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie INDUNI, MD, Study Director — Cabinet dentaire
Locations (2):
- France (2):
  - Cabinet dentaire, Montigny-le-Bretonneux
  - Cabinet dentaire, Paris